CLINICAL TRIAL: NCT06643013
Title: Targeting 18kDa Translocator Protein (TSPO) to Improve Brain Endothelial Cell Function in Cerebral Small Vessel Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24HH8841
Record Dates: First submitted 2024-10-14; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Cerebral Small Vessel Disease
MeSH Terms: conditions — Cerebral Small Vessel Diseases | interventions — N-benzyl-N-ethyl-2-(7,8-dihydro-7-methyl-8-oxo-2-phenyl-9H-purin-9-yl)acetamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XBD173 then Placebo (Experimental)
  Interventions: Drug: XBD173
- Placebo then XBD173 (Experimental)
  Interventions: Drug: XBD173

INTERVENTIONS:
Drug: XBD173 — 4 weeks treatment

SUMMARY:
In healthy people, blood flow to particular areas in the brain increases when the area becomes more active. This ensures that the brain gets enough blood at the right place and time. In people with cerebral small vessel disease (cSVD), this process is disrupted, and the increased blood flow in response to activity is decreased or absent. Damage to the endothelial cells, that form the inner lining of blood vessels, is a key pathological process in cSVD. The aim of this study is to find out whether endothelial cell function and blood flow in cSVD can be improved by altering the function of a protein called TSPO. We will do this by using a drug called XBD173, which binds to TSPO.

This is a double-blind, randomised, crossover study. cSVD patients will be recruited from memory clinics at Imperial College Healthcare NHS Trust. Participants will be invited to the clinical research facility (CRF) at Hammersmith Hospital and randomised to receive XBD173 or matched placebo, twice daily, for 4 weeks. After a 6-week washout, they will be switched to receive the other intervention. The study visits will involve MRI scans and blood tests to assess endothelial cell function.

Healthy volunteers will also be recruited for image optimisation and control data. They will attend for a single MRI scan and not receive XBD173.

ELIGIBILITY:
Inclusion Criteria:

Aged 60-90 years inclusive Male or postmenopausal female

- Men are eligible to participate if they are willing to use the contraception methods listed in the PIS, during treatment and for 90 days after the last dose of treatment Able to provide written informed consent prior to any study-mandated procedures AA genotype at rs6971 (TSPO) locus Imaging-based diagnosis of cSVD (Fazekas score of at least 2 for periventricular and 2 for deep white matter) Mild cognitive impairment (MoCA 18-30) Willing to be genotyped at TSPO and ApoE loci

Inclusion Criteria (Healthy Volunteers):

Aged 60-90 years inclusive Male or female Able to provide written informed consent prior to any study-mandated procedures.

Willing to be genotyped at TSPO and ApoE loci

Exclusion Criteria:

History of clinical stroke History of frequent migraines Known Alzheimer's disease, lewy body disease or evidence of non-vascular neurological diseases Conditions affecting safe engagement in the intervention. Conditions preventing completion of study procedures, e.g. severe loss of vision or hearing Clinically-significant renal disease (eGFR <30 ml/min per 1.73m2) Clinically-significant elevation of serum transaminases or known clinically significant liver disease Contraindications to MRI scanning or exposure to gadolinium-based contrast agents Newly commenced (within 2 months of study start) statins, antihypertensives or antiplatelet treatments Severe respiratory disease with chronic hypoxia (sats <92%), known CO2 retention or need for home oxygen therapy.

Use of the following medications or therapies:

* Severe and moderate P450 CY3A4 inhibitors: Boceprevir, Clarithromycin, Cobicistat, Idelalisib, Itraconazole, Ketoconazole, Nelfinavir, Ritonavir, Saquinavir, Telaprevir, Telithromycin, Voriconazole, Aprepitant, Conivaptan, Crizotinib, Diltiazem, Dronedarone, Erythromycin, Fluconazole, Imatinib, Isavuconazole, Nefazodone, Netupitant, Nilotinib, Posaconazole, Tofisopam, Verapamil, Delavirdine.
* Severe and moderate P450 CY3A4 inducers: Carbamazepine, Enzalutamide, Fosphenytoin, Mitotane, Phenytoin, Rifampicin, Bosentan, Efavirenz, St John's wort, Barbiturates, Nevirapine, Primidone, Rifabutin, Rifapentine.
* Oral contraceptives
* Levothyroxine

Exclusion Criteria (Healthy Volunteers):

Contraindications to MRI scanning or exposure to gadolinium-based contrast agents Pregnant women of childbearing potential Clinically significant renal disease (eGFR <30 ml/min per 1.73m2) Severe respiratory disease with chronic hypoxia (sats <92%), known CO2 retention or need for home oxygen therapy.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Neurovascular coupling | 4 weeks
  Change in primary visual cortex cerebral blood flow following an alertness task

SECONDARY OUTCOMES:
Neurovascular coupling | 4 weeks
  Change in cerebral blood flow in a ROI generated by a group average mask of regions known to become activated in the frontal and temporal lobes
Blood-brain barrier leak | 4 weeks
  BBB leak (rate and volume) determined by gadolinium-enhanced DCE-MRI

OTHER OUTCOMES:
Plasma biomarkers associated with cSVD | 4 weeks
  hsCRP, fibrinogen, IL6, Tnf, TNFR2, osteoprotegerin, VEGF, PGDF, MMP2/9
Plasma biomarkers associated with endothelial cell activation and dysfunction | 4 weeks
  VCAM-1, ICAM-1, E-selectin, von Willebrand factor, plasminogen activator inhibitor-1 activity, soluble ROBO4, VEGF-A, NOS3, tissue plasminogen activator, endothelin-1
Plasma biomarkers of continuing neurodegeneration | 4 weeks
  Neurofilament light chain
Cerebrovascular reactivity in response to CO2 inhalation | 4 weeks
Measure of peripheral endothelial cell function | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul Matthews, PhD, Study Chair — Imperial College London
Locations (1):
- Imperial Clinical Research Facility, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided